CLINICAL TRIAL: NCT04639973
Title: Early Anatomy Scan for Evaluation of Obese Pregnant Women (EASE-O): A Randomized Controlled Trial
Brief Title: Early Anatomy Scan for Evaluation of Obese Pregnant Women (EASE-O)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Cara Buskmiller, Fellow, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HSC-MS-20-0895
Record Dates: First submitted 2020-11-04; First posted 2020-11-23 (Actual); Results first posted 2023-07-13 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: Obesity
Keywords: pregnancy; fetal ultrasound
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group 1 (First trimester ultrasound) (Experimental)
  Interventions: Diagnostic Test: Group 1 (First trimester ultrasound)
- Group 2 (Second trimester anatomy ultrasound) (Active Comparator)
  Interventions: Diagnostic Test: Group 2 (Second trimester anatomy ultrasound)

INTERVENTIONS:
Diagnostic Test: Group 1 (First trimester ultrasound) — A detailed first trimester anatomy ultrasound will be performed,at the visit when the subject is confirmed to be of eligible gestational age. After this detailed research ultrasound, which will be limited to 15 minutes, subject will then receive the clinically indicated dating ultrasound or nuchal translucency measurement. The patient will complete a survey about her satisfaction with this technique via email.as a safety measure, if an anomaly is suspected on the day of the detailed first trimester anatomy scan, the patient will be unblinded. Patients in this arm are later scheduled for a second trimester ultrasound by the clinical team, as this is part of standard obstetrical care.
  Arms: Group 1 (First trimester ultrasound)
Diagnostic Test: Group 2 (Second trimester anatomy ultrasound) — Patients do not undergo a detailed first trimester ultrasound , but will receive the clinically indicated limited ultrasound for dating or for nuchal translucency. Patient will then undergoes a second trimester ultrasound by the clinical team as part of standard obstetrical care and completes a survey regarding her satisfaction with this technique via email.
  Arms: Group 2 (Second trimester anatomy ultrasound)

SUMMARY:
The purpose of this study is to assess the feasibility of ultrasound in the first trimester, assess the completion rate of ultrasounds for fetal anatomy in the first trimester compared to completion rates of ultrasounds for fetal anatomy in the second trimester and to assess the completion rate of the combination of one ultrasound in the first trimester and one in the second trimesters compared to the individual completion rates of both evaluations in obese pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than or equal to 35
* Presented for ultrasound before 14 weeks at The University of Texas Professional Building, Memorial City, Bellaire, or Lyndon-Baines Johnson clinics
* Primary language is English or Spanish
* Consent to an extra transvaginal ultrasound if needed
* Singleton gestation
* No previous anomalies known before consent
* Missed abortion (nonviable pregnancy)

Exclusion Criteria:

* Elective abortion after recruitment
* Missed abortion after first trimester ultrasound
* Did not receive second trimester ultrasound

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cara Buskmiller, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Buskmiller C, Fishel Bartal M, Bonilla M, Denham C, Nguyen R, Sibai B, Pedroza C, Hernandez-Andrade E. First trimester anatomy ultrasound for patients with obesity: a randomized controlled trial. Am J Obstet Gynecol MFM. 2023 Nov;5(11):101143. doi: 10.1016/j.ajogmf.2023.101143. Epub 2023 Sep 3. PMID 37669739
- [Result] Buskmiller C, Toates SE, Rodriguez V, Hernandez-Andrade E. A Learning Curve for First-Trimester Anatomy Ultrasound in Obese Patients. Gynecol Obstet Invest. 2024;89(4):346-350. doi: 10.1159/000538477. Epub 2024 Mar 22. PMID 38522420

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 (First Trimester Ultrasound) | Group 2 (Second Trimester Anatomy Ultrasound)
Started | 65 | 63
Completed | 62 | 62
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Population: Data were not collected from one participant in the group 1 (first trimester ultrasound) arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (First Trimester Ultrasound) | Group 2 (Second Trimester Anatomy Ultrasound) | Total
Number analyzed (Participants) | 64 | 63 | 127
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30.3 [26.3 to 36.6] | 30.9 [27.2 to 34.4] | 30.8 [26.5 to 35.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 63 | 127
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 26 | 51
  Not Hispanic or Latino | 35 | 35 | 70
  Unknown or Not Reported | 4 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21 | 30 | 51
  Black | 30 | 27 | 57
  Asian | 1 | 0 | 1
  Native Hawaiian or Pacific Islander | 10 | 6 | 16
  Other | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 64 | 63 | 127
Insurance [Count of Participants; unit: Participants]
  private | 26 | 21 | 47
  government assisted | 37 | 40 | 77
  self pay | 1 | 1 | 2
  no insurance | 0 | 1 | 1
Marital Status [Count of Participants; unit: Participants]
  Single | 29 | 24 | 53
  Separated | 1 | 1 | 2
  Married | 32 | 34 | 66
  Not Reported | 2 | 4 | 6
Education [Count of Participants; unit: Participants]
  less than highschool | 4 | 1 | 5
  Highschool/GED | 14 | 16 | 30
  some college | 19 | 17 | 36
  college graduate | 12 | 14 | 26
  post graduate | 2 | 5 | 7
  unknown | 13 | 10 | 23
Pre-pregnancy Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 40 [37 to 48] | 40 [38 to 47] | 40 [37.2 to 46.9]
Number of participants with Chronic Hypertension [Count of Participants; unit: Participants] | 18 | 11 | 29
Gestational age at enrollment [Median (Inter-Quartile Range); unit: weeks] | 10.14 [8.57 to 12.14] | 11.00 [8.57 to 12.43] | 10.7 [8.57 to 12.2]
Gestational age at anatomy scan [Median (Inter-Quartile Range); unit: weeks] | 13.3 [13 to 13.7] | 20.4 [20.1 to 21.4] | 18.8 [13.3 to 20.4]
Number of Participants with Type 2 Diabetes Mellitus [Count of Participants; unit: Participants] | 14 | 4 | 18
Parity [Median (Inter-Quartile Range); unit: completed pregnancies] — number of completed pregnancies beyond 20 weeks gestation (whether viable or nonviable)
  completed pregnancies | 1 [0 to 2] | 1 [.5 to 2] | 1 [0 to 2]
Number of Pre-term births [Median (Inter-Quartile Range); unit: pre-term births] — Pre-term birth is defined as babies born alive before 37 weeks of pregnancy are completed.
  pre-term births | 0 [0 to 1] | 0 [0 to 0] | 0 [0 to .25]

OUTCOME MEASURES:

1. Primary Outcome: Completion Rate for First Trimester Scans
Description: Completion rate is reported as the number of scans that see all the views divided by total number of scans in that group
Time Frame: 12-14 weeks of pregnancy
Measure: Number; unit: percent
Arm/Group | Group 1 (First Trimester Ultrasound)
Number analyzed (Participants) | 62
percent | 66

2. Primary Outcome: Completion Rate for Second Trimester Scans
Description: Completion rate is reported as the number of scans that see all the views divided by total number of scans.
Time Frame: 18-22 weeks of pregnancy
Measure: Number; unit: percent
Arm/Group | Group 2 (Second Trimester Anatomy Ultrasound)
Number analyzed (Participants) | 62
percent | 53

3. Secondary Outcome: Completion Rate of First Trimester and Second Trimester Scans
Description: This outcome is reported as [(# of completed 1st tri anatomy scans) + (# of completed 2nd tri anatomy scans in women without a completed first tri anatomy scan)]/(total number of women in first trimester group).
Time Frame: 12-22 weeks of pregnancy
Population: Data was not collected from 62 participants in the Group 2 (second trimester anatomy ultrasound) arm.
Measure: Number; unit: percent
Arm/Group | Group 1 (First Trimester Ultrasound) | Group 2 (Second Trimester Anatomy Ultrasound)
Number analyzed (Participants) | 62 | 0
percent | 82.8 |

4. Secondary Outcome: Time Taken to Complete Scan in the First Trimester Ultrasound Group
Time Frame: 12-14 weeks of pregnancy
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group 1 (First Trimester Ultrasound)
Number analyzed (Participants) | 62
minutes | 65 (27)

5. Secondary Outcome: Number of Anomalies Identified in First Trimester Group Scans
Time Frame: 12-14 weeks of pregnancy
Measure: Number; unit: anomalies
Arm/Group | Group 1 (First Trimester Ultrasound)
Number analyzed (Participants) | 62
anomalies | 5

6. Secondary Outcome: Number of Anomalies Identified in Second Trimester Group Scans
Time Frame: 12-22 weeks of pregnancy
Measure: Number; unit: anomalies
Arm/Group | Group 2 (Second Trimester Anatomy Ultrasound)
Number analyzed (Participants) | 62
anomalies | 6

7. Secondary Outcome: Number of Anomalies Missed in First Trimester Group Scans
Time Frame: 12-14 weeks of pregnancy
Measure: Number; unit: anomalies
Arm/Group | Group 1 (First Trimester Ultrasound)
Number analyzed (Participants) | 62
anomalies | 3

8. Secondary Outcome: Number of Anomalies Missed in Second Trimester Group Scans
Time Frame: 12-22 weeks of pregnancy
Measure: Number; unit: anomalies
Arm/Group | Group 2 (Second Trimester Anatomy Ultrasound)
Number analyzed (Participants) | 62
anomalies | 0

9. Secondary Outcome: Number of Participants With Infants Who Survive
Time Frame: 9 months from randomization
Population: Data was not collected from 4 participants in the Group 1 (first trimester ultrasound) arm.
  Data was not collected from 2 participants in the Group 2 (second trimester anatomy ultrasound) arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (First Trimester Ultrasound) | Group 2 (Second Trimester Anatomy Ultrasound)
Number analyzed (Participants) | 58 | 60
Participants | 57 | 60

10. Secondary Outcome: Gestational Age at Delivery
Time Frame: at the time of delivery (about 40 weeks of pregnancy)
Population: Data was not collected from 5 participants in the Group 1 (first trimester ultrasound) arm.
  Data was not collected from 2 participants in the Group 2 (second trimester anatomy ultrasound) arm.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Group 1 (First Trimester Ultrasound) | Group 2 (Second Trimester Anatomy Ultrasound)
Number analyzed (Participants) | 57 | 60
weeks | 37.4 [34.9 to 38.9] | 37.5 [36.7 to 38.9]

11. Secondary Outcome: Number of Participants With Infants Admitted to the Neonatal Intensive Care Unit (NICU)
Time Frame: at the time of NICU admission (about 0 to 28 days after birth)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (First Trimester Ultrasound) | Group 2 (Second Trimester Anatomy Ultrasound)
Number analyzed (Participants) | 57 | 60
Participants | 18 | 8

12. Secondary Outcome: Hospital Length of Stay
Time Frame: from time of hospital admission to discharge (about 0 to 365 days after birth)
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Group 1 (First Trimester Ultrasound) | Group 2 (Second Trimester Anatomy Ultrasound)
Number analyzed (Participants) | 57 | 60
days | 8 [4.5 to 16.5] | 18 [8.5 to 25.5]

13. Secondary Outcome: Number of Participants With Infants With Neonatal Morbidities
Description: Neonatal morbidities include hypoglycemia
Time Frame: 9 months from randomization
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (First Trimester Ultrasound) | Group 2 (Second Trimester Anatomy Ultrasound)
Number analyzed (Participants) | 57 | 60
Participants | 9 | 3

14. Secondary Outcome: Number of Participants Who Were Very Satisfied With Ultrasound as Measured by the Standardized Survey in the First Trimester Group Scans
Description: The survey asks "Overall, how satisfied were you with today's ultrasound?," and participants selected one of the below choices. Number who chose "Very Satisfied" is reported.
  1. Very satisfied
  2. Somewhat satisfied
  3. Neither satisfied nor dissatisfied
  4. Somewhat dissatisfied
  5. Very dissatisfied
Time Frame: 6 months from randomization
Population: Data was not collected from 32 participants in the Group 1 (first trimester ultrasound) arm. Data was not collected from 62 participants in the Group 2 (second trimester anatomy ultrasound) arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (First Trimester Ultrasound) | Group 2 (Second Trimester Anatomy Ultrasound)
Number analyzed (Participants) | 30 | 0
Participants | 30 |

15. Secondary Outcome: Cost of Intervention Compared to Usual Care
Description: cost benefit analysis based on whether more ultrasounds were done in cases of early discovery of anomalies
Time Frame: from 12-22 weeks of pregnancy
Population: Data were not collected for this outcome measure
Arm/Group | Group 1 (First Trimester Ultrasound) | Group 2 (Second Trimester Anatomy Ultrasound)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From time of enrollment until neonatal discharge from hospital (from about 12 weeks of pregnancy to 365 days after birth)
Description: Data were not collected from one participant in the group 1 (first trimester ultrasound) arm.
Arm/Group | Group 1 (First Trimester Ultrasound) | Group 2 (Second Trimester Anatomy Ultrasound)
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/63
Serious Adverse Events (participants affected / at risk) | 5/64 | 1/63
Other Adverse Events (participants affected / at risk) | 0/64 | 0/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (First Trimester Ultrasound) (N=64) | Group 2 (Second Trimester Anatomy Ultrasound) (N=63)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0)
Fetal death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Neonatal death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT04639973/Prot_SAP_000.pdf